CLINICAL TRIAL: NCT05666856
Title: SBIR Phase II: Scalable Digital Delivery of Evidence-based Training for Family to Maximize Treatment Admission Rates of Opioid Use Disorder in Loved Ones
Brief Title: Scalable Digital Delivery of Evidence-based Training for Family to Maximize Treatment Admission Rates of Opioid Use Disorder in Loved Ones
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: We The Village, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Public Health Management Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2103
Record Dates: First submitted 2022-12-05; First posted 2022-12-28 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-04

CONDITIONS: Community Reinforcement And Family Training; Family Health; Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Conduct a fully-powered RCT comparing two groups. One group will receive digital delivery of the optimized top performing adapted CRAFT intervention from Phase I (CRAFT-A), which consists of a digitally automated curriculum and weekly group coaching sessions, and the second will receive WTV peer support only (PEER).
Who Masked: Outcomes Assessor
Masking Description: The participants will know what group they are in. When data is sent to the statistician for analysis we will code the groups (e.g., 123) without informing which is which. This masks (or blinds) him to the condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRAFT (Experimental): Participants assigned to CRAFT will have access to a 12-module on-line CRAFT intervention and asked to complete one module weekly for 12 weeks. Modules introduce CRAFT concepts and provide workbooks to assist participants in learning and applying the concepts. The modules that are unlocked weekly include: 1) Introduction to CRAFT; 2) Communication Training; 3) Functional Analysis of Drug Using; 4) Positive Reinforcement; 5) Problem-solving; 6) Withdrawing Reinforcement; 7) Allowing Natural Consequences; 8) Life Enrichment; 9) Suggesting Treatment; 10) Recovery and Relapse; 11) Relationship; and 12) Recap of Skills. Two additional modules (domestic violence and opioid overdose precautions) are available at any time. CRAFT participants also attend weekly 60-minute online group sessions facilitated by a CRAFT-certified coach. During weekly group or individual sessions concepts are briefly reviewed, questions are answered, and skills are practiced through role-plays of common situations.
  Interventions: Behavioral: Community Reinforcement And Family Training
- PEER (Active Comparator): Participants assigned to the PEER condition will participate in an online peer support forum with other CSOs. Members of the forum post questions or comments to weekly peer-led discussions and receive responses and feedback from other CSO forum members. Members typically express concerns regarding their IP's wellbeing and ask other members to share any strategies they have employed when dealing with their IPs.
  Interactions typically, are based either in 12-Step strategies members have learned (usually through Al-Anon or Nar-Anon Family Groups or Family Training Workshops provided by treatment programs). A staff member from We The Village monitors forum interactions to ensure members are interacting respectfully.
  Interventions: Behavioral: We The Village Peer Community Forum

INTERVENTIONS:
Behavioral: Community Reinforcement And Family Training — Community Reinforcement Approach and Family Training (CRAFT) is a scientifically based intervention designed to help concerned significant others (CSOs) to engage treatment-refusing substance abusers into treatment. This new intervention method was developed with the belief that the CSO can play a powerful role in helping to engage the substance user in treatment. It is often the substance user who reports that family pressure or influence is the reason sought treatment. CSOs benefit by becoming more independent and reducing their depression, anxiety and anger symptoms even if their loved one does not enter treatment.
  CRAFT uses a positive approach versus confrontation, emphasizing learning new skills to cope with old problems. Some components include: how to stay safe, outlining the context in which substance abusing behavior occurs, teaching CSOs how to use positive reinforcers (rewards) and how to let the substance user suffer the natural consequences for their using behavior.
  Arms: CRAFT
Behavioral: We The Village Peer Community Forum — An online peer support forum with other CSOs. Members of the forum post questions or comments to weekly peer-led discussions and receive responses and feedback from other CSO forum members. Members typically express concerns regarding their IP's wellbeing and ask other members to share any strategies they have employed when dealing with their IPs. Interactions typically, are based either in 12-Step strategies members have learned (usually through Al-Anon or Nar-Anon Family Groups or Family Training Workshops provided by treatment programs) or in CRAFT skills learned (usually from treatment programs or other We The Village members). A staff member from We The Village monitors forum interactions to ensure members are interacting respectfully.
  Arms: PEER

SUMMARY:
The United States is in the midst of an opioid crisis. Over-prescription of opioid analgesic pain relievers contributed to a rapid escalation of use and misuse of these substances across the country. In 2016, more than 2.6 million Americans were diagnosed with opioid use disorder (OUD) and more than 42,000 have died of overdose involving opioids. This death rate is more than any year on record and has quadrupled since 1999 (1,2). Leveraging the potential of available data bases and health IT technologies may help to combat opioid crisis by targeting various aspects of the problem ranging from the prevention of opioid misuse to OUD treatment. NIH through NIDA solicits the research and development of data-driven solutions and services that focus on issues related to opioid use prevention, opioid use, opioid overdose prevention or OUD treatment.

In this project, We The Village, Inc. will address a need to prepare Concerned Significant Others (CSOs) to best use their influence over the trajectory of a loved one's OUD. CSOs are motivated to help, make majority of treatment decisions and payments and have influence over treatment entry and thus, impact the trajectory of an OUD.

The goal of the project is to establish the technical efficacy and commercial viability of CRAFT-A at scale by conducting the fully powered randomized controlled trial (RCT) comparing two online interventions: CRAFT-A (hereinafter referred to as CRAFT or digital CRAFT) and PEER support (the original comparison group). Based on Phase I findings, the team anticipates the CRAFT condition will achieve better outcomes than the PEER condition in a) treatment entry and retention, b) Concerned Significant Others' (CSO) health and wellbeing, c) CSO-IP relationship, and d) CRAFT knowledge.

DETAILED DESCRIPTION:
The primary objective of the proposed Phase II work is to validate technical effectiveness and substantiate commercial viability of delivering CRAFT principles via a data-driven scalable digital program and coaching methods. The Contractor will work with subject matter experts and researchers to achieve the specific aims below.

Technical Objectives 1. Optimize WTV CRAFT-informed prototype and protocol for digital group coaching based on Phase I findings and subject matter advisory input to produce the at-scale prototype.

Technical Objectives 2. Test prototype usability and reliability to deliver the protocol to specifications, and make any refinements needed.

Technical Objectives 3. Demonstrate prototype technical efficacy and commercial viability at scale by conducting a fully powered randomized controlled trial (RCT) comparing two digital interventions: a) CRAFT-A (digitally automated with group coaching), b) PEER support (the original WTV product as a comparison group).

Based on Phase I findings, when tested at baseline versus post-intervention in a randomized clinical trial, the team anticipates the CRAFT-A condition to achieve better outcomes than the PEER condition in a) treatment entry and retention, b) Concerned Significant Others' (CSO) health and wellbeing, c) CSO-IP relationship, and d) CRAFT knowledge. Results will substantiate viability for at scale commercialization and dissemination through WTV's existing and growing network of partners.

ELIGIBILITY:
Inclusion Criteria:

* Is a concerned significant other (CSO) of a loved one with an OUP
* Be 19 years or older
* No substance use disorder
* Has concern about the opioid use of a loved one (IP)
* Plans to be in close contact (phone/face-to-face) with the IP (i.e., 12 days out of 30)
* The IP is not currently receiving treatment, or is in treatment, but the CSO perceives they may benefit from additional treatment (e.g., in residential treatment, but will need to enter outpatient treatment upon discharge or receiving drug free outpatient but not progressing, so may benefit from MAT).

Exclusion Criteria:

* Does not agree to all procedures and sign the consent form
* Is not English-speaking
* Is not able to understand the consent form
* Pass a multiple-choice consent quiz (i.e., 100% correct responses) that tests the participant's comprehension of basic elements of informed consent and the requirements of the protocol administered by the research team over the phone.
* Participants will be given up to three opportunities to pass the consent quiz
* Does not have personal access to a smart phone with data or a computer with internet to be able to access the digital platform for the study conditions, quizzes, questionnaires, and follow-up communication
* Reports that they have a drug abuse problem or a history of drug abuse or dependence and that they have not been in recovery for at least 2 years
* Resides outside the United States
* Participated in previous We The Village pilot study

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-05-04 (Actual); Study Completion 2024-09-22 (Estimated)

PRIMARY OUTCOMES:
New Treatment Entry: IP Treatment Status | 3 months
  Participants report whether their loved one has attended any treatment for their opioid problem since the last assessment by answering 8 questions regarding participation in treatment (e.g., detox, any treatment, new treatment, MAT, new MAT, counseling, support group, and other group). Reports of new treatment, new MAT, and treatment at the follow-up assessment which are not reported at baseline will be categorized as treatment entry. In addition, entry into WTV recovery coaching, WTV family coaching, or reports of treatment entry to WTV staff will be categorized as treatment entry. The outcome is the proportion of participants reporting that their loved one (IP) entered new treatment.

SECONDARY OUTCOMES:
Treatment Retention: IP Treatment Retention Status | 3 months
  Participants report whether their loved one has attended any treatment for their opioid problem since the last assessment by answering 8 questions regarding participation in treatment (e.g., detox, any treatment, new treatment, MAT, new MAT, counseling, support group, and other group). Reports of same treatment, same MAT, and treatment at the follow-up assessment which are reported at baseline will be categorized as treatment retention. In addition, retention in WTV recovery coaching, WTV family coaching, or reports of treatment entry to WTV staff will be categorized as treatment retention. The outcome is the proportion of participants reporting that their loved one (IP) is retained in treatment.
Treatment Retention: IP Treatment Retention Status | 6 months
  Participants report whether their loved one has attended any treatment for their opioid problem since the last assessment by answering 8 questions regarding participation in treatment (e.g., detox, any treatment, new treatment, MAT, new MAT, counseling, support group, and other group). Reports of same treatment, same MAT, and treatment at the follow-up assessment which are reported at baseline will be categorized as treatment retention. In addition, retention in WTV recovery coaching, WTV family coaching, or reports of treatment entry to WTV staff will be categorized as treatment retention. The outcome is the proportion of participants reporting that their loved one (IP) is retained in treatment.
Relationship Happiness: Relationship Happiness Scale | 3 months
  Global score from the 10-item scale was calculated by adding scores (1-10) from 10 items. Minimum possible score was 10 and maximum was 100. Higher scores reflect greater Relationship Happiness.
Relationship Happiness: Relationship Happiness Scale | 6 months
  Global score from the 10-item scale was calculated by adding scores (1-10) from 10 items. Minimum possible score was 10 and maximum was 100. Higher scores reflect greater Relationship Happiness.
CSO Health and Wellbeing: Profile of Mood State (POMS) - Short Form | 3 months
  Total mood disturbance (TMD) score calculated by adding scores (1-5) from the tension (6 items), depression (8 items), anger (7 items), fatigue (5 items), and confusion (5 items) subscales, then subtracting the score form the vigor (6 items) subscale. Minimum TMD possible score was 1 and maximum was 149. Higher scores reflect greater mood disturbance.
CSO Health and Wellbeing: Profile of Mood State (POMS) - Short Form | 6 months
  Total mood disturbance (TMD) score calculated by adding scores (1-5) from the tension (6 items), depression (8 items), anger (7 items), fatigue (5 items), and confusion (5 items) subscales, then subtracting the score form the vigor (6 items) subscale. Minimum TMD possible score was 1 and maximum was 149. Higher scores reflect greater mood disturbance.
CSO Health and Wellbeing: SF-12 Physical Health Subscale | 3 months
  The 7-item scale was transformed so that is had a mean of 50 and a s.d. of 10 in the general US population. Scores above and below 50 are above and below the average with each point representing a difference of 1/10th of a standard deviation.
CSO Health and Wellbeing: SF-12 Physical Health Subscale | 6 months
  The 7-item scale was transformed so that is had a mean of 50 and a s.d. of 10 in the general US population. Scores above and below 50 are above and below the average with each point representing a difference of 1/10th of a standard deviation.
Work Productivity and Activity Impairment: Work Productivity and Activity Impairment questionnaire | 3 months
  The WPAI yeilds four types of scores:
  1. Absenteeism (work time missed)
  2. Presenteesism (impairment at work / reduced on-the-job effectiveness)
  3. Work productivty loss (overall work impairment / absenteeism plus presenteeism)
  4. Activity Impairment WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Work Productivity and Activity Impairment: Work Productivity and Activity Impairment questionnaire | 6 months
  The WPAI yeilds four types of scores:
  1. Absenteeism (work time missed)
  2. Presenteesism (impairment at work / reduced on-the-job effectiveness)
  3. Work productivty loss (overall work impairment / absenteeism plus presenteeism)
  4. Activity Impairment WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
CRAFT Knowledge: CRAFT Knowledge Scale | 3 months
  Measuring the proficiency with which participants answer questions about what to do in scenarios as per the CRAFT approach.
CRAFT Knowledge: CRAFT Knowledge Scale | 6 months
  Measuring the proficiency with which participants answer questions about what to do in scenarios as per the CRAFT approach.
New Treatment Entry: IP Treatment Status | 6 months
  Participants report whether their loved one has attended any treatment for their opioid problem since the last assessment by answering 8 questions regarding participation in treatment (e.g., detox, any treatment, new treatment, MAT, new MAT, counseling, support group, and other group). Reports of new treatment, new MAT, and treatment at the follow-up assessment which are not reported at baseline will be categorized as treatment entry. In addition, entry into WTV recovery coaching, WTV family coaching, or reports of treatment entry to WTV staff will be categorized as treatment entry. The outcome is the proportion of participants reporting that their loved one (IP) entered new treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- We The Village, Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No